CLINICAL TRIAL: NCT07391319
Title: "Prospective, Double-blind, Multicenter, Placebo-controlled, Randomized, Comparative Clinical Study of the Efficacy and Safety of the Drug Neovasculgen® Lyophilisate for the Preparation of a Solution for Intramuscular Administration 1.2 mg", Manufacturer Federal State Budgetary Institution "NMITs of Hematology" of the Ministry of Health of the Russian Federation, Russia in Patients With Diabetic Foot Syndrome"
Brief Title: The Prospective, Double-blind, Multicenter, Placebo-controlled, Randomized, Comparative Clinical Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JSC NextGen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FootDiabEndocrin-05-2024
Record Dates: First submitted 2026-01-12; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ulcer Foot; Mellitus Diabetes
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The investigational therapy group (Neovasculgen) (Experimental): The diluted drug will be administered by 5-10 injections intramuscularly twice with an interval of 14 days, in the course dosage mode - 2.4 mg.
  Interventions: Drug: Neovasculgen®
- The placebo group (Placebo Comparator): Placebo will be administered by 5-10 injections intramuscularly twice with an interval of 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neovasculgen® — The diluted drug will be administered by 5-10 injections intramuscularly twice with an interval of 14 days, in the course dosage mode - 2.4 mg
  Arms: The investigational therapy group (Neovasculgen)
Drug: Placebo — Placebo will be administered by 5-10 injections intramuscularly twice with an interval of 14 days
  Arms: The placebo group

SUMMARY:
The main objective of the study is to evaluate the efficacy and safety of Neovasculgen® in a course dose of 2.4 mg in combination with standard drug therapy in patients with unilateral neuroischemic form of diabetic foot syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years and above inclusive (at the time of study entry) with neuroischemic form of diabetic foot syndrome.
2. Type 1 or type 2 diabetes mellitus.
3. Prolonged non-healing ulcerative defect on the background of standard therapy (at least 1 month), limited to the foot.
4. Depth of ulcer defect according to Wagner Scale- 1 or 2 degrees.
5. Oxygen tension in the tissues directly adjacent to the ulcer defect area, from 20 to 45 mm Hg.
6. Patients with no urgent indications for limb amputation.
7. Acceptable ankle- brachial index range of 1.3-0.25.
8. Patient's willingness to comply with the requirements for examination and treatment.
9. Availability of written informed consent from the patient.
10. Patient's consent to follow the regimen of unloading the affected area throughout the study (for patients with plantar ulcer location)

Exclusion Criteria:

1. Age under 18.
2. Chronic ischemia of the lower limbs of non-atherosclerotic (other than diabetes mellitus) origin: vasculitis, systemic connective tissue diseases, Buerger's disease, congenital anomalies and vascular injuries, embolism.
3. Calcaneal localization of the ulcer.
4. Neuropathic form of diabetic foot syndrome.
5. Severe neuroosteoarthropathic deformity of the foot or other deformity that has a significant impact on the healing process.
6. Ischemia, threatening limb loss.
7. Presence of clinical signs of an infectious process in the ulcer area that is not controlled by the ongoing antibacterial therapy.
8. Presence of purulent-destructive lesions of the foot (abscess, phlegmon, osteomyelitis, etc.).
9. Skin changes associated with venous pathology.
10. Proliferative and terminal stages of diabetic retinopathy.
11. The level of glycated hemoglobin at the entrance to the study is more than 11%.
12. Diabetic ketoacidosis or diabetic precoma.
13. Systemic use of glucocorticosteroids and/or other immunosuppressive drugs within the last 30 days before inclusion in the study.
14. Recent (less than 1 month) surgery or endovascular intervention on the arteries of the lower extremities or recent (less than 1 month) deep vein thrombosis of the lower extremities.
15. Recent (less than 3 months) cases of acute myocardial infarction, unstable angina, coronary artery bypass grafting or stenting of the coronary arteries, stroke or transient ischemic attacks.
16. Planned major surgery in the next 6 months.
17. Severe concomitant disease with life expectancy less than one year.
18. Infectious diseases, septic conditions, HIV infection.
19. Diagnosis of cancer within the last 5 years.
20. Pregnancy, breastfeeding period.
21. Positive pregnancy test in women of reproductive age.
22. Alcohol or drug addiction.
23. Any other disease (including mental) or clinical condition that, in the opinion of the researcher, may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieved complete healing of the ulcer defect through study completion, an average of 6 months | Until the end of the study

SECONDARY OUTCOMES:
Number of participants with partial ulcer defect healing through study completion, an average of 6 months | Until the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Botkin Hospital, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No